CLINICAL TRIAL: NCT04566523
Title: Clinical Benefits of TeleRehabilitation in Chronic Respiratory Failure Patients.
Brief Title: TeleRehabilitation for Patients With Chronic Respiratory Failure.
Acronym: e-mouv
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SOS Oxygene Mediterranee (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-102868-49
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Chronic Respiratory Disease; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Telerehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Chronic respiratory patients who undergo a home-based exercise training program with a rehabilitation coach supervision.
- Tele Group: Chronic respiratory patients who undergo a home-based exercise training program online.
  Interventions: Other: telerehabilitation

INTERVENTIONS:
Other: telerehabilitation — Patients undergo an online exercise training program via a certified host of health data website.
  Groups: Tele Group

SUMMARY:
It is widely described in the literature that exercise training improves patients' exercise tolerance, quality of life, symptoms, anxiety and depression, regardless of the location. Despite overwhelming evidence of the benefits of exercise training, only a very small percentage of eligible people have ever completed a program. Alternative modes of exercise training are needed to improve equity of access for patients with chronic respiratory disease. So TeleRehabilitation, using information and communication technologies to provide distance exercise training services, may be an answer.

ELIGIBILITY:
Inclusion Criteria:

* chronic respiratory disease patients
* Patients with dyspnea or exercise intolerance.
* Stable patients at home.
* Patients who can use a computer (after explanations) and have adequate hearing and vision.
* Collection of the patient's non-objection

Exclusion Criteria:

* Life expectancy <3 months.
* Absolute contraindication to performing physical activity
* Hospitalization for exacerbation in the two months prior to inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from medical consultation
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
exercise tolerance | 3 month after inclusion
  number of steps during 6 minute stepper test

SECONDARY OUTCOMES:
exercise tolerance | 6 month and one year after inclusion
  number of steps during 6 minute stepper test
VQ-11 | 3, 6 month and 1 year after inclusion
  questionnaire, Minimum = 11, maximum = 55; higher score means worth outcome
physical activity quantity | 3, 6 month and 1 year after inclusion
  questioning patients on their physical activity quantity

CONTACTS AND LOCATIONS:
Overall Officials: william Heurtaux, MD, Principal Investigator — Clinique des Cèdres
Locations (1):
- Cabinet de pneumologie Clinique des Cèdres, Cornebarrieu, France

IPD SHARING:
Plan to Share IPD: No